CLINICAL TRIAL: NCT07095166
Title: Monitoring Eating Across Locations (MEAL) - Timing, Intake, and Mealtime Evaluation (TIME)
Acronym: MEAL-TIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Alaina Pearce, PI, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00026981
Record Dates: First submitted 2025-07-09; First posted 2025-07-31 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Obesity
Keywords: eating behavior; meal microstructure; child; obesity
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home than Lab Meal (Experimental): Participant is randomly assigned to eat the study meal at home first and then in the lab
  Interventions: Behavioral: Meal Location
- Lab then Home Meal (Experimental): The participant receives the study meal in the Lab first and then at Hoem
  Interventions: Behavioral: Meal Location

INTERVENTIONS:
Behavioral: Meal Location — The location at which the child will eat the experimental meal - home or lab

SUMMARY:
Increased availability of high-energy dense foods has contributed to a pediatric obesity epidemic, with 23% of United States children currently presenting with the disease. How children eat contributes to both overconsumption and greater adiposity. However, it is unclear if laboratory measures of children's eating style generalize to the home environment, where children consume two thirds of their total energy. The study will 1) test if child eating styles observed in the lab generalize to more ecologically valid home environments and 2) identify aspects of home food environment that amplify obesogenic eating behaviors. We will assess laboratory and home eating styles (e.g., bite rate) in 100 prepubertal 6-9-year-old children to constrain variability in energy requirements. Children will be video-recorded while consuming identical study-provided meals at home and in the laboratory (counter-balanced order) in addition to a 'typical' meal at home. To study how adiposity relates to "obesogenic" styles of eating, gold standard dual x-ray absorptiometry will be used.

ELIGIBILITY:
Inclusion Criteria:

* children must be between the ages of 6-9 years-old
* children are of good health with no learning disabilities (e.g., ADHD, determined by parent report)
* children are not on any medications known to impact body weight, taste, food intake, behavior, or blood flow
* parents report that children like and are willing to eat study foods

Exclusion Criteria:

* they are not within the age requirements (<6 years old or > 9 years old)
* If they are taking cold or allergy medication, or other medications known to influence cognitive function, taste, appetite, or blood flow.
* If they don't speak English.
* If they are colorblind.
* If they have a learning disability, ADD/ADHD, language delays, autism or other neurological or psychological conditions.
* If they have a pre-existing medical condition such as type I or type II diabetes, rheumatoid arthritis, Cushing's syndrome, Down's syndrome, severe lactose intolerance, Prader-Willi syndrome, HIV, cancer, renal failure, or cerebral palsy.
* If they are allergic to foods or ingredients used in the study.
* child received an X-ray in the previous year (to avoid excess radiation exposure due to the DXA scans performed in the research)

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Child body mass index | Day 1
  child height and weight will be measured
Food intake in grams during a standard meal | Day 1 and Day 2 or 3 depending on randomization
  Intake in grams from standard meal
Food intake in kcal during a standard meal | Day 1 and Day 2 or 3 depending on randomization
  Intake in kcal during a standard meal
Video coding of standard meal | Day 1 and Day 2 or 3 depending on randomization
  A digital recording of the child eating a standard meal will be saved. We have developed a behavior coding protocol to measure child meal microstructure (e.g., bites, bite size, meal duration). We have also validated a computational model to assess cumulative intake curves from video coded bite data.
Food intake in grams during a snack buffet when not hungry | Day 1
  Intake in grams during a snack buffet using a standard eating in the absence of hunger paradigm (i.e., non-homeostatic intake)
Food intake in kcal during a snack buffet when not hungry | Day 1
  Intake in kcal during a snack buffet using a standard eating in the absence of hunger paradigm (i.e., non-homeostatic intake)
Body Composition | Day 1
  Dual-energy X-ray absorptiometry to assess body composition including fat mass and fat-free mass in children
Food intake in grams during a Study Meal | Day 2 or 3 depending on randomization and home meal administration
  Intake in grams from Study Meal
Food intake in kcal during the Study Meal | Day 2 or 3 depending on randomization and home meal administration
  Intake in kcal during the Study Meal
Video coding of the study meal | Day 2 or 3 depending on randomization and home meal administration
  ! digital recording of the child eating a Study Meal will be saved. We have developed a behavior coding protocol to measure child meal microstructure (e.g., bites, bite size, meal duration). We have also validated a computational model to assess cumulative intake curves from video coded bite data.
Video coding of home meals | Week 1 and Week 2
  Digital recordings of the child eating a typical meals at home. We have developed a behavior coding protocol to measure child meal microstructure (e.g., bites, bite size, meal duration). We have also validated a computational model to assess cumulative intake curves from video coded bite data.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD will be shared. For identifiable video data, data will only be shared if participants consent to sharing their videos in a restricted repository called Databrary.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD will be available at the end of the study and be available in perpetuity
Access Criteria: De-identified IPD will be openly available while identifiable IPD will be available through a restricted access repository called Databrary. identifiable data shared with Databrary will only be viewable and downloadable to authorized users who have been granted secure access by Databrary's administrators. Only researchers with Principal Investigator status from institutions with Institutional Review Boards or similar review entities, or researchers affiliated with Principal Investigators, will be authorized for access.
  Authorized users will be required to sign a user agreement that specifies that they will: (1) be responsible for maintaining the confidentiality of the data; (2) abide by ethical principles for treatment of human subjects as mandated by their local Institutional Review Boards; (3) agree not use the data for commercial purposes; and (4) treat data in Databrary with the same high standards of care that they would treat data collected in their own laboratories.

REFERENCES:
- [Background] Neuwald NV, Pearce AL, Cunningham PM, Setzenfand MN, Koczwara L, Rolls BJ, Keller KL. Food switching at a meal is positively associated with change in adiposity among children at high-familial risk for obesity. Appetite. 2025 Apr 1;208:107915. doi: 10.1016/j.appet.2025.107915. Epub 2025 Feb 25. PMID 40010570
- [Background] Neuwald NV, Pearce AL, Adise S, Rolls BJ, Keller KL. Switching between foods: A potential behavioral phenotype of hedonic hunger and increased obesity risk in children. Physiol Behav. 2023 Oct 15;270:114312. doi: 10.1016/j.physbeh.2023.114312. Epub 2023 Aug 4. PMID 37543104
- [Background] Fogel A, Fries LR, McCrickerd K, Goh AT, Quah PL, Chan MJ, Toh JY, Chong YS, Tan KH, Yap F, Shek LP, Meaney MJ, Broekman BFP, Lee YS, Godfrey KM, Fong Chong MF, Forde CG. Oral processing behaviours that promote children's energy intake are associated with parent-reported appetitive traits: Results from the GUSTO cohort. Appetite. 2018 Jul 1;126:8-15. doi: 10.1016/j.appet.2018.03.011. Epub 2018 Mar 15. PMID 29551400
- [Background] Fogel A, Goh AT, Fries LR, Sadananthan SA, Velan SS, Michael N, Tint MT, Fortier MV, Chan MJ, Toh JY, Chong YS, Tan KH, Yap F, Shek LP, Meaney MJ, Broekman BFP, Lee YS, Godfrey KM, Chong MFF, Forde CG. A description of an 'obesogenic' eating style that promotes higher energy intake and is associated with greater adiposity in 4.5year-old children: Results from the GUSTO cohort. Physiol Behav. 2017 Jul 1;176:107-116. doi: 10.1016/j.physbeh.2017.02.013. Epub 2017 Feb 14. PMID 28213204
- [Background] Fogel A, Goh AT, Fries LR, Sadananthan SA, Velan SS, Michael N, Tint MT, Fortier MV, Chan MJ, Toh JY, Chong YS, Tan KH, Yap F, Shek LP, Meaney MJ, Broekman BFP, Lee YS, Godfrey KM, Chong MFF, Forde CG. Faster eating rates are associated with higher energy intakes during an ad libitum meal, higher BMI and greater adiposity among 4.5-year-old children: results from the Growing Up in Singapore Towards Healthy Outcomes (GUSTO) cohort. Br J Nutr. 2017 Apr;117(7):1042-1051. doi: 10.1017/S0007114517000848. Epub 2017 May 2. PMID 28462734
- [Background] Pearce AL, Cevallos MC, Romano O, Daoud E, Keller KL. Child meal microstructure and eating behaviors: A systematic review. Appetite. 2022 Jan 1;168:105752. doi: 10.1016/j.appet.2021.105752. Epub 2021 Oct 16. PMID 34662600
- [Background] Pearce AL, Adise S, Roberts NJ, White C, Geier CF, Keller KL. Individual differences in the influence of taste and health impact successful dietary self-control: A mouse tracking food choice study in children. Physiol Behav. 2020 Sep 1;223:112990. doi: 10.1016/j.physbeh.2020.112990. Epub 2020 Jun 4. PMID 32505786